CLINICAL TRIAL: NCT07237269
Title: Abiraterone/Prednisone + Standard ADT vs Standard ADT for Prostate Cancer Patients With PSMA-Positive Conventional Imaging Negative Pelvic Lymphadenopathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 787-25-FB
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard ADT (Active Comparator): Standard Hormone Therapy
  Interventions: Drug: Hormone therapy
- Abiraterone/Prednisone + Standard ADT (Experimental): Abiraterone/Prednisone Combination plus Standard Hormone Therapy
  Interventions: Drug: Hormone therapy

INTERVENTIONS:
Drug: Hormone therapy — Abiraterone/Prednisone + Standard Hormone Therapy (ADT) = Enhanced Hormone Therapy; Standard Hormone Therapy (ADT) alone = SOC

SUMMARY:
The advent of PSMA-PET has allowed greater sensitivity and specificity when staging prostate cancers, particularly intermediate and high-risk prostate cancers. This has created a gap in knowledge regarding the treatment of patients who have PSMA-positive but conventionally negative pelvic lymphadenopathy (i.e. <1cm in smallest diameter). The purpose of this study is to compare outcomes of enhanced ADT with abiraterone and prednisone and standard ADT, both alongside radiation therapy, in prostate cancer patients with PSMA-positive but conventionally negative pelvic lymphadenopathy. We hypothesize that enhanced ADT with abiraterone and prednisone is superior to standard ADT for the treatment of prostate cancer patients with PSMA-positive but conventionally negative pelvic lymphadenopathy. We further hypothesize that standard ADT will be associated with a lower rate of adverse events. 140 eligible patients will be randomized to receive either enhanced ADT with abiraterone and prednisone or standard ADT, both with concurrent radiation therapy. Patients will be followed for 5 years after completion of ADT to evaluate outcomes. The primary objective will be to determine if enhanced ADT has superior 5-year failure-free survival compared to standard ADT. Secondary objectives include evaluation of chronic toxicities, quality of life impact, biochemical progression-free survival, cancer-specific survival, overall survival, and metastasis-free survival. Additionally, the study will have two exploratory objectives involving assessment of tumor growth rate and regression rate using PSA values and determine the correlation of treatment efficacy and toxicity with blood-based Heme oxygenase 1 (HO-1) concentration. If enhanced ADT is not superior to standard ADT for prostate cancer patients with PSMA-positive but conventionally negative pelvic lymphadenopathy, this would suggest that treatment with standard ADT may be adequate and thus be a strong impetus for larger multi-institutional clinical trials to investigate this notion.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven diagnosis of local prostate cancer. Biopsies will be confirmed by UNMC pathology review if collected outside our institution.
2. Targetable PSMA-avid pelvic lymph node measuring <1cm in short axis diameter.
3. No prior definitive treatment or intervention received.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 within 14 days prior to registration.
5. Age ≥ 30 years.
6. Patient must be able to provide study-specific informed consent prior to study entry.
7. Patient must be able to swallow medications.

Exclusion Criteria:

1. Evidence of distant metastatic disease outside the pelvic lymph nodes (including osseous pelvic disease).
2. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse.
3. Relative or absolute contraindications to radiation therapy as determined by the treating physician. These include, but are not limited to, inflammatory bowel disease, connective tissue disorders (systemic lupus erythematosus, scleroderma, etc.), and genetic disorders that risk increased sensitivity to radiation therapy.
4. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 3 months prior to registration.
   2. Congestive heart failure (NYHA functional capacity class II or greater).
   3. Transmural myocardial infarction within the last 3 months prior to registration.
   4. History of stroke or transient ischemic attack within 3 months prior to registration.
   5. Currently uncontrolled diabetes mellitus.
   6. Ongoing arrhythmias of Grade >2 [National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE), version 5.03]; chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
   7. Thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism) in the past month.
   8. Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
   9. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
   10. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
   11. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
   12. Acquired Immune Deficiency Syndrome (AIDS) based upon the current Centers for Disease Control and Prevention definition that is being treated with contraindicated medications, including but not limited to Atazanavir, Saquinavir, Ritonavir, Indinavir, or Nelfinavir. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   13. Uncontrolled seizures or seizures in the past 3 months. Patients can enroll if their seizures have been well-controlled for >3 months on antiseizure medications.
   14. Gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE version 5 grade 3 or greater within 30 days prior to registration.
   15. History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to registration.
   16. Total bilirubin ≥1.5X upper limit of normal (ULN) [except for subjects with Gilbert's disease, in which case total bilirubin not to exceed 10X ULN], alanine (ALT) and aspartate (AST) aminotransferase >= 2.5X ULN.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
5-year failure-free survival rate | 7 years
  Determine the impact of enhanced ADT with abiraterone/prednisone versus standard ADT on the 5-year failure-free survival of patients with PSMA-positive conventionally negative pelvic lymphadenopathy (i.e. <1cm in smallest diameter).

SECONDARY OUTCOMES:
Toxicity in both arms from 3 months to 2 years post-ADT. | 4-years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Evaluate and compare patient-reported symptom outcomes in both arms from 3 months to 2 years post-ADT. (IPSS) | 4-years
  Using IPSS (International Prostate Symptom Score). The quality of life measures will be summarized using descriptive statistics at each time point collected as n, mean, SD, median, minimum, and maximum.
Evaluate and compare patient-reported symptom outcomes in both arms from 3 months to 2 years post-ADT. (FACT-P) | 4-years
  Using FACT-P (Functional Assessment of Cancer Therapy-Prostate.) The quality of life measures will be summarized using descriptive statistics at each time point collected as n, mean, SD, median, minimum, and maximum.
Evaluate local progression-free survival (i.e., failure-free survival excluding biochemical failure). | 7-Years
  Evaluate progression-free survival (i.e., failure-free survival excluding biochemical failure). Progression-free survival will be estimated with the Kaplan-Meier method and will be compared between treatment arms with the log-rank test. The 5-year survival rates will be estimated with a 95% confidence interval. Time to local failure is defined as time since randomization to disease progression within the intact prostate. Regional, metastases, and deaths are treated as competing events.
Evaluate locoregional progression-free survival (i.e., failure-free survival excluding biochemical failure). | 7-Years
  Evaluate progression-free survival (i.e., failure-free survival excluding biochemical failure). Progression-free survival will be estimated with the Kaplan-Meier method and will be compared between treatment arms with the log-rank test. The 5-year survival rates will be estimated with a 95% confidence interval.
  Time to locoregional failure is defined as time since randomization to disease progression within the pelvis and pelvic lymph nodes. Metastases and deaths are treated as competing events.
Evaluate 5-year overall survival | 7-Years
  Overall survival will be estimated with the Kaplan-Meier method and will be compared between treatment arms with the log-rank test. The 5-year survival rates will be estimated with a 95% confidence interval. Overall survival is defined as the time since the date of randomization to the date of death or last follow-up.
Evaluate 5-year cancer-specific survival | 7-Years
  Cumulative incidence methods will be used to estimate 5-year rates (with 95% CI) of LC, LRC, and DM while accounting for death as a competing event. Cancer-specific survival is defined as time since the date of randomization to the date of death due to cancer diagnosis or treatment or last follow-up. Deaths due to other causes are treated as competing events.
Evaluate 5-year metastasis-free survival. | 7-Years
  Time to distant metastasis is defined as time since date of randomization to distant metastases in para-aortic lymph nodes and distant organs or last follow-up. Locoregional failures and deaths are treated as competing events.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share